CLINICAL TRIAL: NCT03605160
Title: Efficacy of Fluid-jet as an Innovative Method to Prevent Posterior Capsular Opacity After Phacoemulsification
Brief Title: An Innovative Method Fluid-jet to to Remove Residual Lens Fibers
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Haotian Lin, professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CCPMOH2018-China-5
Record Dates: First submitted 2018-07-06; First posted 2018-07-30 (Actual); Last update posted 2019-05-29 (Actual); Status verified 2019-05

CONDITIONS: Posterior Capsule Opacification
Keywords: cataract surgery; polish; residual lens fibers; fluid-jet

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- traditional group (Active Comparator): Perform conventional continuous curvilinear capsulorhexis. After phacoemulsification and I/A, switch to polish mode and use I/A instrument to remove the RLFs visible on the posterior capsule before injection of viscoelastic agent. IOP: 55mmHg; Aspiration: 0-10; Vacuum: 0-20. The standard for stopping polish is that the RLFs can no longer be absorbed by the side holes on the I/A instrument in this mode, or there are no discernible RLFs on the posterior capsule. If RLFs on the posterior capsular are found after IOL implantation, polish to remove them after the removal of viscoelastic agents. All operations are videotaped during the whole operation. The total polish time is recorded as the time of all polish procedures.
  Interventions: Procedure: traditional polish
- fluid-jet group (Experimental): Perform conventional continuous curvilinear capsulorhexis. After phacoemulsification and I/A, inject viscoelastic agent and implant IOL without polish. Use I/A instrument to remove viscoelastic agent. A 27G irrigating syringe was used, and the RLFs on the posterior capsule were gently aligned to make a fluid-jet basically parallel to the iris. The liquid pressure of 50-120 mmHg is produced. The standard for stopping in this mode is that the RLFs can no longer be washed down from the capsule, or there are no discernible RLFs on the posterior capsule. All operations are videotaped during the whole operation. The total time of all jet procedures recorded in the videotape is the total time of jet.
  Interventions: Procedure: fluid-jet

INTERVENTIONS:
Procedure: traditional polish — After phacoemulsification and I/A, switch to polish mode and use I/A instrument to remove the RLFs visible on the posterior capsule before injection of viscoelastic agent. IOP: 55mmHg; Aspiration: 0-10; Vacuum: 0-20. The standard for stopping polish is that the RLFs can no longer be absorbed by the side holes on the I/A instrument in this mode, or there are no discernible RLFs on the posterior capsule. If RLFs on the posterior capsular are found after IOL implantation, polish to remove them after the removal of viscoelastic agents.
  Arms: traditional group
Procedure: fluid-jet — After phacoemulsification and I/A, inject viscoelastic agent and implant IOL without polish. Use I/A instrument to remove viscoelastic agent. A 27G irrigating syringe was used, and the RLFs on the posterior capsule were gently aligned to make a fluid-jet basically parallel to the iris. The liquid pressure of 50-120 mmHg is produced. The standard for stopping in this mode is that the RLFs can no longer be washed down from the capsule, or there are no discernible RLFs on the posterior capsule.
  Arms: fluid-jet group

SUMMARY:
Residual lens fibers (RLFs) on the posterior lens capsule during cataract surgery can cause after cataract, affecting visual quality and increasing the medical cost for further laser posterior capsulotomy. However, conventional polish is inconvenient and time-consuming. We use an innovative fluid-jet method to remove RLFs, and compare the efficacy of fluid-jet and polish to prevent posterior capsular opacity after phacoemulsification.

DETAILED DESCRIPTION:
Purpose: Residual lens fibers (RLFs) on the posterior lens capsule during cataract surgery can cause after cataract, affecting visual quality and increasing the medical cost for further laser posterior capsulotomy. However, conventional polish is inconvenient and time-consuming. We use an innovative fluid-jet method to remove RLFs, and compare the efficacy of fluid-jet and polish to prevent posterior capsular opacity after phacoemulsification.

Design: Single-center, prospective, randomized controlled clinical study Subjects of study: Age-related cataract patients receiving phacoemulsification from Zhongshan Ophthalmic Center, Guangzhou, China.

Methods: patients are 1: 1 randomized to two groups. Polish group: After irrigation and aspiration (I/A), the RLFs on the posterior capsule are removed by polishing before intraocular lens (IOL) implantation; Fluid-jet group: Polish is not performed. RLFs on posterior capsule are removed by jetting fluid with an irrigating syringe after IOL implantation. The posterior capsular images of all the patients are obtained immediately before and after IOL implantation, and at the end of surgery, then the amount of RLFs is quantitatively analyzed by using LYZ-PCO, a software we developed. Best corrected visual acuity and parameters of visual quality, such as objective scattering index(OSI), Strehl ratio (SR) and Modulation Transfer Function (Mtf)-cut off are evaluated by objective visual quality analyser (OQAS) at 1 day, 1 week and 1 year after surgery. The patients receives telephone follow-up every month. The severity of posterior capsular opacification (PCO) and incidence of laser posterior capsulotomy is recorded.

Main indicators for the study: The incidence of laser posterior capsulotomy a year after surgery.

ELIGIBILITY:
Iinclusion criteria:

1) cataract patients aged between 50 and 80 years; 2) graded 5 or less for lens opalescence by the Lens Opacities Classification System, version III (LOCS III); 3) listed for phacoemulsification combined with intraocular lens implantation in topical anesthesia; 4) Signed informed consent.

Exclusion criteria:

1) a history ophthalmic trauma or surgery; 2) other ophthalmic diseases such as glaucoma, uveitis, high myopia; 3) diabetes requiring medical control; 4) disagree with follow-up monitoring; 5) Other factors inappropriate to participate in this project, including but not limited to severe cataracts, very shallow anterior chambers, etc.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 740 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2023-01-01 (Estimated); Study Completion 2023-01-01 (Estimated)

PRIMARY OUTCOMES:
change in rate of posterior capsulotomy | 1 year, 2 year, 3 year, 4 year, 5 year after surgery
  Incidence rate of laser posterior capsulotomy

SECONDARY OUTCOMES:
change in visual acuity | 1 day, 1 week, 1 year post-op, and every year thereafter.
  Best corrected visual acuity tested with ETDRS chart
change in objective scattering index | 1 day, 1 week, 1 year post-op, and every year thereafter.
  objective scattering index of participants
change in Strehl ratio | 1 day, 1 week, 1 year post-op, and every year thereafter.
  Strehl ratio of participants
change in modulation transfer function cut off | 1 day, 1 week, 1 year post-op, and every year thereafter.
  Modulation transfer function cut off of participants
area of posterior capsular opacification | 1 year, 2 year, 3 year, 4 year, 5 year after surgery
  posterior capsular opacification area percentage
residual lens fibers | the amount of residual lens fibers is to be measured for every participant using ocular image taken with surgical microscope at the end of the cataract surgery
  amount of residual lens fibers at the posterior lens capsule

CONTACTS AND LOCATIONS:
Overall Officials: Yizhi Liu, M.D., Ph.D., Study Chair — Zhongshan Ophthalmic Center, Sun Yat-sen University
Locations (1):
- Zhognshan Ophthalmic Center, Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No